CLINICAL TRIAL: NCT07154979
Title: Effective Dose of Oliceridine for Inhibiting Hemodynamic Elevation Induced by Tracheal Intubation: An Up-and-Down Sequential Trial
Brief Title: Oliceridine Dose for Tracheal Intubation Hemodynamic Elevation: Up-and-Down Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiyou Wei (Other)
Responsible Party: Sponsor-Investigator, Shiyou Wei, Department of Anesthesiology, Shanghai Pulmonary Hospital, Shanghai, China
Organization: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20250250
Record Dates: First submitted 2025-08-06; First posted 2025-09-04 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-09

CONDITIONS: Oliceridine
Keywords: oliceridine; dose-finding; µ-opioid receptor G-protein-biased agonist; up-and-down sequential design
MeSH Terms: interventions — ((3-methoxythiophen-2-yl)methyl)((2-(9-(pyridin-2-yl)-6-oxaspiro(4.5)decan-9-yl)ethyl))amine

STUDY DESIGN:
Intervention Model Description: A single-group, up-and-down sequential dose-finding design to determine the ED₅₀ and ED₉₅ of oliceridine for suppression of hemodynamic responses to tracheal intubation.
Masking Description: Open-label study; participants, investigators, and outcome assessors are aware of the intervention assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oliceridine Up-and-Down Sequential Dose-Finding Arm (Experimental): In this single-group, up-and-down sequential design, adult patients receive a single intravenous bolus of oliceridine.
  * Initial dose: 45 µg/kg for ages 18-65 years; 40 µg/kg for ≥ 65 years
  * Two minutes later: propofol 2 mg/kg iv
  * At loss of consciousness (MOAA/S ≤ 1): rocuronium 0.6 mg/kg iv
  * Direct-laryngoscope tracheal intubation performed upon full muscle relaxation
  * Hemodynamic variables (BP, HR) recorded at baseline, 2 min post-oliceridine, immediately pre-intubation, and for 3 min post-intubation
  * A "positive" response (hemodynamic surge) is defined as ≥ 20% increase in MAP or HR, HR ≥ 120 bpm, or SBP ≥ 180 mmHg
  * Next patient's oliceridine dose is adjusted ± 3 µg/kg according to the preceding patient's response
  * Sequential dosing continues until seven crossovers are observed, allowing estimation of ED₅₀ and ED₉₅.
  Interventions: Drug: Oliceridine Injection

INTERVENTIONS:
Drug: Oliceridine Injection — Adult participants receive a single IV bolus of oliceridine (initial dose 45 µg/kg for ages 18-65 y or 40 µg/kg for ≥65 y). Two minutes later, propofol 2 mg/kg IV is administered. Upon loss of consciousness (MOAA/S ≤ 1), rocuronium 0.6 mg/kg IV is given. Direct laryngoscopic tracheal intubation is performed after full muscle relaxation. Blood pressure and heart rate are recorded at baseline, 2 min post-oliceridine, immediately pre-intubation, and for 3 min post-intubation. A "positive" hemodynamic response is defined as ≥ 20% increase in MAP or HR, HR ≥ 120 bpm, or SBP ≥ 180 mmHg. Subsequent oliceridine doses are adjusted ± 3 µg/kg based on the prior patient's response until seven response crossovers are observed, allowing estimation of ED₅₀ and ED₉₅.
  Other Names: TRV130

SUMMARY:
This is a clinical trial using an up-and-down sequential design, aiming to investigate the median effective dose (ED50) and 95% effective dose (ED95) of oliceridine for inhibiting hyperdynamic responses induced by tracheal intubation during general anesthesia induction. The study will enroll patients undergoing elective tracheal intubation under general anesthesia, stratified into young (18-65 years) and elderly (≥65 years) groups. By dynamically adjusting oliceridine doses, the optimal induction dose in different age groups will be evaluated to provide reference for rational clinical medication.

DETAILED DESCRIPTION:
1. Study Objectives To determine the ED50 and ED95 of oliceridine in inhibiting tracheal intubation-induced hyperdynamic responses (e.g., increased blood pressure and heart rate) during general anesthesia induction, and to provide dose evidence for individualized anesthesia induction protocols.
2. Study Design Type: A dynamic dose-finding clinical trial using the modified Dixon up-and-down sequential design.

   Sample Size: 35 cases per group anticipated, with trial termination after 7 cross-overs between positive and negative responses (i.e., transitions in whether hemodynamic responses exceed 20% of baseline).

   Grouping: Stratified by age into young group (18-65 years) and elderly group (≥65 years).
3. Study Participants

   Inclusion Criteria:

   Patients undergoing elective tracheal intubation under general anesthesia; Aged ≥18 years; American Society of Anesthesiologists (ASA) physical status Ⅰ-Ⅲ; Body mass index (BMI) < 25.

   Exclusion Criteria:

   Systolic blood pressure (SBP) ≥160 mmHg, diastolic blood pressure (DBP) ≥110 mmHg, or heart rate ≥110 beats/min at rest upon admission to the operating room; Long-term use of analgesics or sedatives before surgery; Pregnancy, lactation, or planned pregnancy; Allergy to oliceridine; Mental illness or inability to communicate normally.
4. Trial Procedures Screening Period (-7 to 0 days): Informed consent signed; collection of basic information (age, ASA class, etc.); baseline blood pressure and heart rate monitored.

   Anesthesia Induction and Intubation:

   Routine vital sign monitoring and intravenous access established upon patient admission.

   Initial doses: 45 μg/kg for the young group and 42 μg/kg for the elderly group. Subsequent doses adjusted based on intubation response (increase by 3 μg/kg for positive response, decrease by 3 μg/kg for negative response).

   Administration sequence: Intravenous oliceridine → propofol 2 mg/kg 2 minutes later → rocuronium 0.6 mg/kg after loss of consciousness (MOAA/S score ≤1) → tracheal intubation after neuromuscular blockade.

   Anesthesia Maintenance: Propofol (4-8 mg/kg/h) and remifentanil (0.05-0.1 μg/kg/min) infused continuously; rocuronium added intermittently; protective ventilation strategy applied.
5. Outcome Measures Primary Measures: ED50 and ED95 of oliceridine for inhibiting post-intubation hyperdynamic responses.

   Secondary Measures:

   Incidence of hyperdynamic responses within 3 minutes after intubation; Blood pressure (SBP, DBP) and heart rate at baseline, 2 minutes after drug administration, before intubation, and within 3 minutes after intubation; Modified Observer's Assessment of Alertness/Sedation (MOAA/S) score; Adverse events (arrhythmia, coughing, allergic reactions, etc.).
6. Statistical Methods Data analysis will be performed using R software. Quantitative data will be expressed as mean±standard deviation or median (interquartile range), and qualitative data as frequency (percentage). Probit analysis will be used to calculate ED50 and its 95% confidence interval. A P-value <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery requiring general anesthesia with tracheal intubation
* Age ≥ 18 years
* American Society of Anesthesiologists (ASA) physical status I-III
* BMI<25

Exclusion Criteria:

* At rest in the operating room, systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 110 mmHg or heart rate ≥ 110 bpm
* Preoperative long-term use of analgesic or sedative medications
* Pregnancy, breastfeeding, known or planned pregnancy
* Known allergy or hypersensitivity to oliceridine or any study medication components
* History of psychiatric illness or inability to communicate effectively

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2025-09-04 (Actual); Primary Completion 2025-09-11 (Actual); Study Completion 2025-09-11 (Actual)

PRIMARY OUTCOMES:
ED₉₅ of oliceridine for suppression of tracheal intubation-induced hemodynamic response | From the start of intubation to 3 minutes after the end of intubation
  95% effective dose (ED₉₅) of oliceridine required to prevent a positive hemodynamic response-defined as ≥ 20% increase in mean arterial pressure or heart rate, heart rate ≥ 120 bpm, or systolic blood pressure ≥ 180 mmHg-within 3 minutes after tracheal intubation during general anesthesia induction, estimated by probit regression analysis of up-and-down sequential dosing data.
ED₅₀ of oliceridine for suppression of tracheal intubation-induced hemodynamic response | From the start of intubation to 3 minutes after the end of intubation
  Median effective dose (ED₅₀) of oliceridine required to prevent a positive hemodynamic response-defined as ≥ 20% increase in mean arterial pressure or heart rate, heart rate ≥ 120 bpm, or systolic blood pressure ≥ 180 mmHg-within 3 minutes after tracheal intubation during general anesthesia induction, estimated by probit regression analysis of up-and-down sequential dosing data.

SECONDARY OUTCOMES:
The number of cases with coughing | From the start of anesthesia induction to 3 minutes after the end of intubation
  During anesthesia induction, intravenous injection of opioids may cause coughing. During the intubation process, coughing may occur due to airway stimulation.

OTHER OUTCOMES:
Changes in blood pressure at predefined time points | From baseline through 3 minutes after tracheal intubation.
  Systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP) are recorded at:
  Baseline (prior to oliceridine administration) 2 minutes after oliceridine bolus Immediately before tracheal intubation The highest values within 3 minutes following intubation
The number of cases with adverse events | up to 1 day after surgery
  Including arrhythmia (abnormal heart rhythms such as tachycardia, arrhythmia, etc.), body movement (involuntary limb movements during anesthesia induction and intubation), airway spasm (airway narrowing caused by contraction of airway smooth muscles, accompanied by dyspnea, wheezing, etc.), allergic reaction (allergic responses induced by trial drugs or other anesthetics, such as rash, pruritus, hypotension, etc.), as well as patient-reported symptoms like palpitation (sensation of abnormal heartbeat) and dyspnea (labored breathing, abnormal respiratory rate, or insufficient ventilation)
Success rate of sedation | From the start of intubation to 3 minutes after the end of intubation
  The modified observer's assessment of alert/sedation scale (MOAA/S) is a commonly - used sedation evaluation tool in clinical practice. It classifies reactivity under different stimuli: Grade 5 means a sensitive response to calling the name in a normal tone of voice; Grade 4 indicates a sluggish response to calling the name in a normal tone of voice; Grade 3 requires a loud or repeated call of the name to elicit a response; Grade 2 shows a response to slight pushing and vibration; Grade 1 has a response to a painful stimulus (by squeezing the trapezius muscle area); Grade 0 means no response to a painful stimulus. Moreover, MOAA/S ≤ 2 indicates loss of consciousness, which can assist medical staff in judging the sedation level and consciousness state of patients.
Heart rate at predefined time points | From baseline through 3 minutes after tracheal intubation.
  Heart rate (HR) are recorded at:
  Baseline (prior to oliceridine administration) 2 minutes after oliceridine bolus Immediately before tracheal intubation The highest values within 3 minutes following intubation

CONTACTS AND LOCATIONS:
Overall Officials: Shiyou Wei, PhD, Study Chair — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Tianmen First People's Hospital, Tianmen, Hubei, China

IPD SHARING:
Plan to Share IPD: No